# Ceftazidime-avibactam plasma levels in critically ill patients, including those receiving continuous renal replacement therapy

# NCT04358991

# SIGNATURE PAGE

# **RESPONSIBLE STUDY AUTHORS**

| STUDY AUTHOR(S): |
|---|
| I have read this report and confirm that to the best of my knowledge it accurately describes the conduct and results of the study. |
| Signature: Date: _April 7, 2020 |
| Ryan K. Shields |
| Principal Investigator |
| University of Pittsburgh |
| 3550 Terrace Street, Room S805 |
| Pittsburgh, PA 15621 |

412-864-3745

# **Table of Contents**

| SIGNATURE PAGE | 1 |
|---|---|
| RESPONSIBLE STUDY AUTHORS | 1 |
| Table of Figures. | 3 |
| Table of Tables. | 3 |
| List of Abbreviations. | 4 |
| Purpose5 | |
| Methods 5 | |
| Results7 | |
| Ceftazidime Pharmacokinetics | 9 |
| Avibactam Pharmacokinetics | 11 |
| Pharmacokinetic Parameters: Patients Receiving Renally-Adjusted Doses of CAZ-AVI | 13 |
| Pharmacodynamics and Target Attainment | 15 |
| Safety | 16 |
| References | |
| Appendix | 1818 |

# Table of Figures.

| Figure 1. Chromatograms of Ceftazidime and Avibactam | 6 |
|---|---|
| Figure 2. Ceftazidime Plasma Concentrations in Patients Receiving 2.5g IV q 8h | 9 |
| Figure 3. Ceftazidime Concentration-time Profile: Patients Receiving 2.5g IV q 8h, Stratified by those with | n or |
| without CRRT | 10 |
| Figure 4. Avibactam Plasma Concentrations in Patients Receiving 2.5g IV q 8h | 11 |
| Figure 5. Avibactam Concentration-time Profile: Patients Receiving 2.5g IV q 8h, Stratified by those with | |
| without CRRT | 12 |
| Figure 6: Concentration-time profiles of Patients Receiving Non-standard Dosing | 14 |
| Figure 7. Target Attainment for Ceftazidime. | 15 |
| Figure 8. Target Attainment for Avibactam | 16 |
| Table of Tables. | |
| Table 1. Patient Demographics (n=20) | 7 |
| Table 2. Renal Replacement Therapy Settings. | 8 |
| Table 3. Calculated Ceftazidime PK parameters by Patient Group | |
| Table 4. Ceftazidime PK Parameters for Patients Receiving Continuous Renal Replacement Therapy | |
| Table 5. Calculated Avibactam PK Parameters by Patient Group. | 11 |
| Table 6. Avibactam PK Parameters for Patients Receiving Continuous Renal Replacement Therapy | |
| Table 7. Measured Total Drug Values of Ceftazidime and Avibactam in Critically III Patients. | |

### List of Abbreviations.

AUC - area under curve

AVI – avibactam

CAZ – ceftazidime

CL – observed clearance at steady state

CLSI - Clinical and Laboratory Standards Institute

cm - centimeter

C<sub>max</sub> – predicted maximum concentration

C<sub>min</sub> – predicted minimum concentration

CrCI - creatinine clearance

CRRT – continuous renal replacement therapy

CVVHDF - continuous venovenous hemodiafiltration

EDTA – ethylenediaminetetraacetic acid

*f*T – time of free drug concentration

g – gram

HD - hemodialysis

IBW – ideal body weight

IQR - interquartile range

IV – intravenous(ly)

K<sub>e</sub> – equilibrium constant

kg - kilogram

LCMS - liquid chromatography mass spectrometry

MIC – minimum inhibitory concentration

µg/mL – micrograms per millilter

PD – pharmacodynamics

PK – pharmacokinetic

RRT – renal replacement therapy

q 8/24/48h - every 8/24/48 hours

t<sub>1/2</sub> – half life

UHPLC – ultra high performance liquid chromatography

V<sub>d</sub> – observed volume of distribution at steady state

### Purpose.

Ceftazidime-avibactam is a  $\beta$ -lactam/ $\beta$ -lactamase inhibitor combination used to treat multidrug-resistant gramnegative infections. There are limited pharmacokinetic data among critically ill patients and no dosing recommendations for those receiving continuous renal replacement therapy (CRRT). The objective of this study is to describe the population pharmacokinetics of ceftazidime and avibactam among patients infected or being treated for multidrug-resistant gram-negative pathogens, including those on CRRT.

### Methods.

### **Enrollment**

Adult patients at UPMC Presbyterian hospital who received >24 hours of ceftazidime-avibactam were eligible for participation. Informed consent was obtained for each subject. The study protocol was approved by the University of Pittsburgh institutional review board (protocol number: PRO17060377).

### **Clinical management**

During the course of the study, we identified receipt of RRT as a risk factor for clinical failure and emergence of ceftazidime-avibactam resistance [1]. Given these data, our standard approach to ceftazidime-avibactam treatment for patients receiving CRRT was to administer 2.5g IV q 8h and enroll patients into this study. For each of these patients, we carefully monitored patients for any signs or symptoms of drug toxicity, including neurotoxicity and myelosuppression.

### Sampling and storage

Whole blood samples were collected from November 2016 to March 2019 in sterile tubes containing EDTA as an anticoagulant. Samples were collected prior to a dose of ceftazidime-avibactam, and then at 2, 4, 6, and 8 hours after the infusion started. Collection tubes were centrifuged at 3,000 x rpm for 5 minutes immediately after collection. Plasma was stored in 0.5-1mL aliquots at -80°C until analysis.

# Simultaneous measurement of avibactam and ceftazidime with a highly-sensitive, reproducible ultra high performance liquid chromatography mass spectrometry (UHPLC-MS) assay.

We developed an UHPLC-MS assay to quantify avibactam and ceftazidime on a Shimadzu Nexera XD UHPLC with a Shimadzu 8045 MS (Figure 1). Mobile phase A was 0.1% formic acid in water; mobile phase B was 0.1% formic acid in acetonitrile. Samples were prepared by adding 100 $\mu$ L of plasma to 200 $\mu$ L of water and 700 $\mu$ L of acetonitrile containing internal standards (ceftazidime-d5, Toronto Research Chemical, Toronto Canada; avibactam-H2; Alsachim, Illkirch, France). Samples were vortexed, allowed to rest on ice, then centrifuged at 13,000 x rpm for 5 minutes, and allowed to rest on ice again. In an LCMS vial, 100 $\mu$ L of supernatant was added to 400 $\mu$ L mobile phase A and samples were loaded into a 4°C autosampler. A Waters Atlantis T3 column (3 $\mu$ m, 50x2.1mm; with guard) was used. An elution gradient at 0.5mL/min started at 5% B increasing to 90% B, where it was held for 30 seconds before returning to 5% B. The total run time was 5.5 minutes and the injection volume was 3 $\mu$ L. Transitions were monitored in positive mode for ceftazidime (m/z 274.1 < 80.05) and negative mode for avibactam (264.00 < 95.90). The assay was reproducible and linear over a range of 0.1 - 20 $\mu$ g/mL for avibactam and 1 - 200 $\mu$ g/mL for ceftazidime.



Figure 1. Chromatograms of Ceftazidime and Avibactam.

## Pharmacokinetic and Pharmacodynamic analysis.

Pharmacokinetic analysis of serum concentrations was performed with WinNonlin version 8.2 (Certara, Princeton, NJ) for IV infusion noncompartmental model analysis. Predicted PK values were calculated for each patient. Descriptive statistics are provided, including mean and standard deviation for continuous variables. Dichotomous or continuous variables were compared by chi-squared test or Mann-Whitney U, respectively.

### Results.

A total of 20 patients (Table 1) were enrolled in the study. Fifteen patients received a standard dosing regimen of 2.5g ceftazidime-avibactam every 8 hours intravenously. Five patients received dose-adjustments due to renal insufficiency. Two received 1.25g of ceftazidime-avibactam every 8 hours intravenously, 2 received 0.94g every 48 hours, and 1 received 0.94g every 24 hours. For patients receiving CRRT, dialysis settings and flow rates are provided in Table 2.

Table 1. Patient Demographics (n=20).

| Patient # | Age | Sex | Race <sup>1</sup> | Height<br>(cm) | Weight <sup>2</sup><br>(kg) | Dose | SCr on day of sampling | Cockroft-<br>Gault IBW<br>(kg) | Renal<br>Replacement<br>Therapy |
|---|---|---|---|---|---|---|---|---|---|
| 7 | 74 | F | D | 160 | 50.9 | 0.94g q 24h | 2.3 | CRRT | CRRT |
| 2 | 64 | М | W | 178 | 66 | 0.94g q 48h | 2 | HD | HD |
| 5 | 69 | F | W | 173 | 54.5 | 0.94g q 48h | 2.1 | HD | HD |
| 1 | 60 | М | W | 185 | 120.8 | 1.25g q 8h | 2.1 | 42.0 | None |
| 16 | 51 | F | W | 168 | 65.7 | 1.25g q 8h | 1.5 | 42.0 | None |
| Mean (non-standard dosing): | 63.6 | | | 172.8 | 71.6 | | 1.93 | | |
| 3 | 59 | F | W | 163 | 70.1 | 2.5g q 8h | 1 | 52.6 | None |
| 4 | 59 | F | W | 163 | 78.2 | 2.5g q 8h | 0.6 | 87.7 | None |
| 6 | 59 | F | W | 185 | 85.8 | 2.5g q 8h | 0.7 | 133.5 | None |
| 8 | 66 | M | W | 175 | 132 | 2.5g q 8h | 0.4 | CRRT | CRRT |
| 9 | 68 | М | W | 175 | 75.6 | 2.5g q 8h | 1.2 | CRRT | CRRT |
| 10 | 48 | F | W | 173 | 67 | 2.5g q 8h | 1.5 | CRRT | CRRT |
| 11 | 35 | M | W | 163 | 66 | 2.5g q 8h | 1 | CRRT | CRRT |
| 12 | 59 | М | U | 170 | 120 | 2.5g q 8h | 1.5 | CRRT | CRRT |
| 13 | 58 | М | W | 178 | 96 | 2.5g q 8h | 1.5 | CRRT | CRRT |
| 14 | 45 | F | W | 163 | 46.2 | 2.5g q 8h | 0.4 | 154.2 | None |
| 15 | 44 | F | W | 168 | 132 | 2.5g q 8h | 0.4 | 168.6 | None |
| 17 | 31 | М | W | 193 | 75.5 | 2.5g q 8h | 0.7 | 187.1 | None |
| 18 | 61 | М | W | 168 | 104.6 | 2.5g q 8h | 1 | 70.2 | None |
| 19 | 41 | М | W | 171 | 73.2 | 2.5g q 8h | 2.5 | 36.8 | None |
| 20 | 63 | М | W | 177 | 114 | 2.5g q 8h | 0.8 | 96.3 | None |
| Mean (standard dosing): | 53.1 | | | 172.3 | 89.0 | | 1.01 | | |
| Mean (overall): | 55.7 | | | 172.4 | 84.7 | | 1.21 | | |

<sup>&</sup>lt;sup>1</sup>White (W), declined race (D), race unknown (U)

<sup>&</sup>lt;sup>2</sup>Adjusted body weight was used for obese patients when >120% IBW

Table 2. Renal Replacement Therapy Settings.

| Patient | CRRT<br>Machine | Type of CRRT | Filter Model | Blood Flow Rate<br>(mL/hr) | Replacement Fluid<br>Infusion Rate<br>(mL/hr) | Dialysate Flow Rate<br>(mL/hr) |
|---|---|---|---|---|---|---|
| 7 | Prismaflex | CVVHDF | M100 | 250 | 250 | 1750 |
| 8 | Prismaflex | CVVHDF | M100 | 250 | 250 | 3000 |
| 9 | Prismaflex | CVVHDF | M100 | 200 | 500 | 2000 |
| 10 | Prismaflex | CVVHDF | M100 | 250 | 250 | 1500 |
| 11 | Prismaflex | CVVHDF | M100 | 250 | 250 | 1700 |
| 12 | Prismaflex | CVVHDF | M150 | 300 | 250 | 3500 |
| 13 | Prismaflex | CVVHDF | M100 | 250 | 250 | 2500 |

### **Ceftazidime Pharmacokinetics**

A total of 96 plasma samples were collected from 20 patients. Figure 2 shows total ceftazidime concentrations plotted for each patient. Table 3 lists PK parameters for all patients stratified by dosing strategy. There was no statistical difference (Mann-Whitney) between patients receiving a standard 2.5g dose q8h with normal renal function and patients on CRRT for  $C_{max}$ , AUC, CL, and  $V_d$ . Median values were statistically different for  $C_{min}$  (normal function 29.01 vs CRRT 46.59, p = 0.0496), t<sub>1/2</sub> (normal function 4.478h vs CRRT 10.12h, p = 0.0496), and the rate elimination constant ( $K_e$ ) (normal function 0.15 vs CRRT 0.07, p = 0.0496). Figure 3 compares the concentrations over time per patient for those with and without CRRT.

Figure 2. Ceftazidime Plasma Concentrations in Patients Receiving 2.5g IV q 8h.



Table 3. Calculated Ceftazidime PK parameters by Patient Group.

| Median | All patients | | Othor (1975) | | | |
|---|---|---|---|---|---|---|
| (IQR) | (n=20) | All 2.5g q8h<br>(n=15) | CrCl > 50ml/min<br>(n=9); 2.5g IV q8h | CRRT (n=6);<br>2.5g IV q8h | <i>P</i> value | Other (n=5) |
| C <sub>max</sub> (µg/ml) | 80.6 (61.2,<br>104.1) | 87.0 (69.2, 108.2) | 81.3 (76.5, 88.1) | 96.3 (69.6,<br>112.4) | 0.4559 | 69.9 (59.3, 73.2) <sup>1</sup> |
| C <sub>min</sub> (µg/mI) | 40.4 (28.3, 55.0) | 35.4 (27.7, 53.5) | 29.0 (20.9, 35.5) | 46.6 (37.9, 64.4) | 0.0496 | 46.1 (46.0, 53.7) <sup>1</sup> |
| AUC <sub>0-8h</sub><br>(hr*µg/mL) <sup>2</sup> | 456.3 (400.3<br>588.1) | 456.6 (388.7,<br>651.8) | 437.4 (328.2,<br>550.3) | 522.2 (455.1,<br>683.7) | 0.3277 | 444.8 (432.7, 456.9) |
| K <sub>e</sub> (1/hr) | 0.13 (0.06, 0.16) | 0.15 (0.10, 0.16) | 0.15 (0.14, 0.19) | 0.07 (0.05, 0.14) | 0.0496 | 0.04 (0.04, 0.07) |
| t <sub>1/2</sub> (hr) | 5.2 (4.3, 12.6) | 4.5 (4.2, 7.0) | 4.5 (3.7, 5.1) | 10.1 (5.5, 15.1) | 0.0496 | 15.7 (8.9, 16.5) |
| V <sub>d</sub> (L) | 34.6 (22.5, 49.3) | 28.7 (20.6, 46.0) | 26.0 (16.3, 36.1) | 43.2 (31.3, 56.9) | 0.1135 | 40.7 (33.1, 55.1) |
| CL (L) | 3.6 (2.3, 5.2) | 4.4 (3.2, 5.5) | 5.3 (3.6, 6.2) | 4.0 (3.0, 4.7) | 0.2238 | 2.3 (1.8, 2.3) |

<sup>&</sup>lt;sup>1</sup> See Table 6 for details.

 $<sup>^{2}</sup>$  For AUC, patients with 24 or 48 hour dosing were excluded; All patients n = 17, Other n = 2

Figure 3. Ceftazidime Concentration-time Profile: Patients Receiving 2.5g IV q 8h, Stratified by those with or without CRRT.



Table 4. Ceftazidime PK Parameters for Patients Receiving Continuous Renal Replacement Therapy.

| Patient | Regimen | C <sub>min</sub><br>(µg/ml) | C <sub>max</sub><br>(µg/ml) | AUC <sub>0-8h</sub><br>(hr*μg/mL) | t <sub>1/2</sub><br>(hr) | CL<br>(L/hr) | V <sub>d</sub><br>(L) | Blood<br>Flow<br>Rate<br>(mL/hr) | Replacement<br>Fluid Infusion<br>Rate (mL/hr) | Dialysate<br>Flow Rate<br>(mL/hr) |
|---|---|---|---|---|---|---|---|---|---|---|
| 8 | 2.5g IV q 8h | 45.73 | 60.43 | 456.3 | 16.24 | 5.92 | 143.92 | 250 | 250 | 3000 |
| 9 | 2.5g IV q 8h | 22.72 | 104.95 | 454.7 | 4.32 | 5.54 | 34.43 | 200 | 500 | 2000 |
| 10 | 2.5g IV q 8h | 80.03 | 162.85 | 1156.4 | 16.77 | 2.18 | 53.24 | 250 | 250 | 1500 |
| 11 | 2.5g IV q 8h | 45.88 | 83.33 | 588.1 | 4.40 | 4.45 | 30.40 | 250 | 250 | 1700 |
| 12 | 2.5g IV q 8h | 30.85 | 70.91 | 377.1 | 8.60 | 6.46 | 76.61 | 300 | 250 | 3500 |
| 13 | 2.5g IV q 8h | 68.26 | 122.98 | 715.6 | 11.64 | 3.48 | 54.80 | 250 | 250 | 2500 |

### **Avibactam Pharmacokinetics**

The same 96 samples were simultaneously analyzed for avibactam total drug concentrations; Figure 4 shows the results for each patient. Table 5 lists PK parameters for all patient groups. There was no statistical difference (Mann-Whitney) between patients receiving a standard 2.5g dose q8h with normal renal function and patients on CRRT for  $C_{max}$  or  $V_d$ . Median values for  $C_{min}$ , AUC,  $t_{1/2}$ ,  $K_e$ , and CL were statistically different (normal function vs CRRT, respectively: 4.45 vs 11.1, p = 0.0028, 73.4 vs 126.4, p = 0.0496, 3.3 vs 10.3, p = 0.0048, 0.21 vs 0.07, p = 0.0048, 6.6 vs 4.2, p = 0.0256). Figure 5 shows the time course results for the 15 standard dose patients.

Figure 4. Avibactam Plasma Concentrations in Patients Receiving 2.5g IV q 8h.



Table 5. Calculated Avibactam PK Parameters by Patient Group.

| Median | All patients | | Othor (25) | | | |
|---|---|---|---|---|---|---|
| (IQR) | (n=20) | All 2.5g q8h<br>(n=15) | CrCl > 50ml/min<br>(n=9); 2.5g IV q8h | CRRT (n=6); 2.5g<br>IV q8h | P value | Other (n=5) |
| C <sub>max</sub><br>(µg/ml) | 15.6 (11.8, 23.0) | 15.9 (12.7, 24.3) | 13.3 (11.3, 16.3) | 21.3 (16.7, 27.1) | 0.1135 | 14.1 (8.9,<br>21.5) <sup>1</sup> |
| C <sub>min</sub><br>(µg/ml) | 8.5 (4.2, 9.8) | 8.9 (3.9, 10.1) | 4.5 (2.8, 8.9) | 11.1 (9.8, 14.2) | 0.0028 | 6.11 (5.8, 9.0) <sup>1</sup> |
| AUC <sub>0-8h</sub><br>(hr*µg/mL) <sup>2</sup> | 98.8 (58.3, 149.4) | 99.1 (62.0, 150.2) | 73.4 (48.3, 99.1) | 126.4 (101.9,<br>154.5) | 0.0496 | 74.7 (66.5,<br>82.9) |
| K <sub>e</sub> (1/hr) | 0.15 (0.07, 0.21) | 0.16 (0.09, 0.21) | 0.21 (0.16, 0.23) | 0.07 (0.05, 0.13) | 0.1135 | 0.07 (0.05,<br>0.07) |
| t <sub>1/2</sub> (hr) | 4.6 (3.3, 10.2) | 4.4 (3.3, 7.9) | 3.3 (3.0, 4.2) | 10.3 (5.6, 15.2) | 0.0048 | 9.8 (9.3, 12.6) |
| V <sub>d</sub> (L) | 43.2 (23.4, 58.9) | 38.1 (22.6, 56.8) | 32.1 (20.6, 43.8) | 56.1 (35.4, 78.9) | 0.1135 | 43.8 (42.6,<br>57.7) |
| CL (L) | 4.5 (3.3, 6.2) | 5.3 (3.4, 8.0) | 6.6 (5.6, 9.6) | 4.2 (3.3, 4.9) | 0.0256 | 3.0 (1.6, 3.6) |

<sup>&</sup>lt;sup>1</sup> See Table 6 for details.

<sup>&</sup>lt;sup>2</sup> For AUC, patients with 24 or 48 hour dosing were excluded; All patients n = 17, Other n = 2

Figure 5. Avibactam Concentration-time Profile: Patients Receiving 2.5g IV q 8h, Stratified by those with or without CRRT.



Table 6. Avibactam PK Parameters for Patients Receiving Continuous Renal Replacement Therapy.

| Patient | Regimen | C <sub>min</sub><br>(µg/ml) | C <sub>max</sub><br>(µg/ml) | AUC <sub>0-8h</sub><br>(hr*μg/mL) | t <sub>1/2</sub><br>(hr) | CL<br>(L/hr) | V <sub>d</sub><br>(L) | Blood<br>Flow<br>Rate<br>(mL/hr) | Replacement<br>Fluid Infusion<br>Rate (mL/hr) | Dialysate<br>Flow Rate<br>(mL/hr) |
|---|---|---|---|---|---|---|---|---|---|---|
| 8 | 2.5g IV q 8h | 10.11 | 13.43 | 101.4 | 16.36 | 5.33 | 130.64 | 250 | 250 | 3000 |
| 9 | 2.5g IV q 8h | 5.04 | 23.79 | 103.4 | 4.35 | 4.87 | 30.64 | 200 | 500 | 2000 |
| 10 | 2.5g IV q 8h | 20.28 | 38.15 | 279.5 | 31.83 | 1.79 | 84.40 | 250 | 250 | 1500 |
| 11 | 2.5g IV q 8h | 11.66 | 20.74 | 149.4 | 4.52 | 3.49 | 24.26 | 250 | 250 | 1700 |
| 12 | 2.5g IV q 8h | 8.26 | 17.97 | 98.8 | 8.94 | 4.97 | 62.56 | 300 | 250 | 3500 |
| 13 | 2.5g IV q 8h | 14.66 | 28.12 | 156.2 | 11.66 | 3.17 | 49.66 | 250 | 250 | 2500 |

# Pharmacokinetic Parameters: Patients Receiving Renally-Adjusted Doses of CAZ-AVI.

Five patients received non-standard dosing. Table 7 details the dose received, as well as the observed concentrations of both ceftazidime and avibactam at specific times following start of drug infusion. Figure 6 show the concentration-time profiles of these patients for both ceftazidime (top panels) and avibactam (bottom panels).

Table 7. Measured Total Drug Values of Ceftazidime and Avibactam in Critically III Patients.

| Patient | Dosing | Creatinine<br>clearance or RRT | Actual Draw Time<br>(hours) <sup>1</sup> | Ceftazidime<br>(µg/mL) | Avibactam<br>(μg/mL) |
|---|---|---|---|---|---|
| | | | Pre-dose | 38.563 | 8.692 |
| | | | 2.1 | 76.049 | 17.473 |
| 7 | 0.94g IV q 24h | CRRT | 3.3 | 66.048 | 16.391 |
| | | | 6.1 | 58.712 | 14.380 |
| | | | 7.4 | 55.094 | 13.026 |
| | 2. 0.94g IV q 48h | | Pre-dose | 4.436 | 1.056 |
| 2 | | HD <sup>2</sup> | 14.5 (Pre-HD) | 18.848 | 4.643 |
| 2 | 0.94917 4 4011 | | 16.5 (Mid-HD) | 8.385 | 1.845 |
| | | | 18.4 (Post-HD) | 4.790 | 1.069 |
| | | | 2.4 (Pre-HD) | 23.864 | 7.583 |
| 5 | 0.94g IV q 48h | HD <sup>3</sup> | 5.9 (Post-HD) | 7.049 | 1.721 |
| 3 | 0.94917 4 4011 | TID | 24.8 | 7.742 | 2.265 |
| | | | 48.1 | 6.925 | 2.099 |
| | | | 4.2 | 61.665 | 11.960 |
| 1 | 1.25g IV q 8h | 42mL/min | 6.1 | 52.092 | 10.208 |
| | | | 7.9 | 46.306 | 9.071 |
| 16 | 1.25g IV q 8h | 42mL/min | 2.0 | 59.388 | 8.903 |
| 10 | 1.20917 4 011 | 721112/111111 | 5.3 | 51.557 | 7.009 |

<sup>&</sup>lt;sup>1</sup>Time relative to start of drug infusion.

<sup>&</sup>lt;sup>2</sup> Patient received a full 4-hour HD session with 1L ultrafiltration. Samples were collected immediately before, during, and after HD.

<sup>&</sup>lt;sup>3</sup> Patient received a 3-hour HD session with 1.5L ultrafiltration. Samples were collected immediately before and after HD, as well as 24 and 48 hours after the dose. The latter time point represents the trough values for this patient.

Figure 6: Concentration-time profiles of Patients Receiving Non-standard Dosing.



### **Pharmacodynamics and Target Attainment**

Ceftazidime free drug concentration was calculated by adjusting for 10% protein binding. To determine if patients in the study met pre-determined PD targets, we assessed the time free drug concentrations (*f*T) remained above the MIC and 4x MIC, using the CLSI susceptibility breakpoint for ceftazidime (8 µg/mL) as the representative MIC value. All patients dosed every 8 hours had ceftazidime exposures of 100% *f*T>MIC (Figure 7). Both patients receiving intermittent dialysis achieved targets before, but not after HD. Excluding patients on HD, 56% of patients achieved exposures of 100% *f*T>4xMIC, an exposure reported to suppress the emergence of resistance [2].



Figure 7. Target Attainment for Ceftazidime.

For analysis purposes, we estimated the avibactam free drug concentration using 10% protein binding as well [3]. Although PD targets are not as well elucidated for  $\beta$ -lactamase inhibitors, we used surrogate targets of 1 and 2.5  $\mu$ g/mL and evaluated free trough concentrations of avibactam. As shown in Figure 8, 95% and 90% of patients met targets of 100% fT>1  $\mu$ g/mL and >2.5  $\mu$ g/mL, respectively [2-4]. Only one patient (patient #17) with normal function on a standard 2.5g g8h dose did not meet targets.

Figure 8. Target Attainment for Avibactam.



## Safety

The safety of ceftazidime-avibactam has been well-defined for patients with normal renal clearance, but not for patients receiving standard doses during CRRT. We assessed 6 such patients as part of this study to ensure exposures, which clearly met PD targets, were not associated with undue toxicity. Among the 6 patients receiving 2.5g IV q 8h on CRRT (Table 2), 50% died within 72 hours of sample collection due to underlying multi-system organ failure. One additional patient was transitioned to HD the day after study enrollment. The last two patients received treatment courses of 12 and 14 days with no apparent toxicity, including myelosuppression, neurotoxicity, or further renal toxicity.

#### References.

- 1. Shields, R.K., et al., *Pneumonia and Renal Replacement Therapy Are Risk Factors for Ceftazidime-Avibactam Treatment Failures and Resistance among Patients with Carbapenem-Resistant Enterobacteriaceae Infections*. Antimicrob Agents Chemother, 2018. **62**(5).
- 2. Li, J., et al., Ceftazidime-Avibactam Population Pharmacokinetic Modeling and Pharmacodynamic Target Attainment Across Adult Indications and Patient Subgroups. Clin Transl Sci, 2019. **12**(2): p. 151-163.
- 3. Sy, S.K.B., et al., Clinical Pharmacokinetics and Pharmacodynamics of Ceftazidime-Avibactam Combination: A Model-Informed Strategy for its Clinical Development. Clin Pharmacokinet, 2019. **58**(5): p. 545-564.
- 4. Shields, R. and Y. Doi, *Aztreonam Combination Therapy: A Long-Awaited Answer to Metallo-beta-Lactamase-Producing Gram-Negatives?* Clin Infect Dis, 2019.
- 5. Soukup, P., et al., Steady-State Ceftazidime-Avibactam Serum Concentrations and Dosing Recommendations in a Critically III Patient Being Treated for Pseudomonas aeruginosa Pneumonia and Undergoing Continuous Venovenous Hemodiafiltration. Pharmacotherapy, 2019. **39**(12): p. 1216-1222.
- 6. Wenzler, E., et al., *Pharmacokinetics and Dialytic Clearance of Ceftazidime-Avibactam in a Critically III*Patient on Continuous Venovenous Hemofiltration. Antimicrob Agents Chemother, 2017. **61**(7).
- 7. Veillette, J.J., J. Truong, and S.C. Forland, *Pharmacokinetics of Ceftazidime-Avibactam in Two Patients With KPC-Producing Klebsiella pneumoniae Bacteremia and Renal Impairment.* Pharmacotherapy, 2016. **36**(11): p. e172-e177.
- 8. Nicolau, D.P., et al., *Phase 1 study assessing the steady-state concentration of ceftazidime and avibactam in plasma and epithelial lining fluid following two dosing regimens*. J Antimicrob Chemother, 2015. **70**(10): p. 2862-9.
- 9. Stein, G.E., et al., *Pharmacokinetic and Pharmacodynamic Analysis of Ceftazidime/Avibactam in Critically III Patients*. Surg Infect (Larchmt), 2019. **20**(1): p. 55-61.

# Appendix.

Observed Drug Concentrations.

| Patient | # hours post start of infusion | Total Measured CAZ (μg/mL) | Total Measured AVI (μg/mL) |
|---|---|---|---|
| 1 | 4.22 | 61.665 | 11.960 |
| | 6.08 | 52.092 | 10.208 |
| | 7.92 | 46.306 | 9.071 |
| 2 | -2.28 | 4.436 | 1.056 |
| | 14.50 | 18.848 | 4.643 |
| | 16.50 | 8.385 | 1.845 |
| | 18.42 | 4.790 | 1.069 |
| 3 | -0.70 | 69.076 | 12.027 |
| | 2.47 | 149.718 | 29.957 |
| | 4.02 | 114.670 | 20.922 |
| | 5.85 | 87.003 | 14.256 |
| | 8.15 | 57.749 | 8.816 |
| 4 | 1.05 | 114.512 | 19.102 |
| | 2.13 | 124.009 | 19.293 |
| | 4.13 | 59.349 | 6.936 |
| | 5.63 | 46.217 | 4.894 |
| | 6.13 | 40.060 | 4.245 |
| | 8.63 | 25.943 | 2.461 |
| | -0.25 | 26.280 | 2.302 |
| 5 | 2.42 | 23.864 | 7.583 |
| | 5.92 | 7.049 | 1.721 |
| | 24.83 | 7.742 | 2.265 |
| | 29.20 | 8.935 | 2.596 |
| | 48.07 | 6.925 | 2.099 |
| 6 | 2.33 | 71.190 | 12.212 |
| | 4.45 | 36.178 | 4.575 |
| | 6.40 | 27.501 | 3.054 |
| | 7.28 | 23.193 | 2.521 |
| 7 | -0.12 | 38.563 | 8.692 |
| | 2.05 | 76.049 | 17.473 |
| | 3.30 | 66.048 | 16.391 |
| | 6.13 | 58.712 | 14.380 |
| | 7.35 | 55.094 | 13.026 |
| 8 | 0.05 | 45.727 | 10.111 |
| | 2.55 | 60.427 | 13.428 |
| | 6.30 | 49.106 | 10.919 |
| | 8.58 | 47.102 | 10.487 |
| 9 | -0.17 | 22.724 | 5.042 |
| | 2.45 | 104.953 | 23.793 |
| | 3.03 | 78.604 | 17.805 |

| | 3.93 | 60.631 | 13.852 |
|----|-------|---------|--------|
| | 5.98 | 41.508 | 9.548 |
| | 7.97 | 31.745 | 7.291 |
| 10 | -0.18 | 80.026 | 20.284 |
| | 0.85 | 140.574 | 33.392 |
| | 1.98 | 162.853 | 38.147 |
| | 3.87 | 156.434 | 36.869 |
| | 6.00 | 138.158 | 34.962 |
| 11 | 0.00 | 53.859 | 14.073 |
| | 1.12 | 83.329 | 20.740 |
| | 2.47 | 75.611 | 19.423 |
| | 4.17 | 82.851 | 20.739 |
| | 6.08 | 63.154 | 16.557 |
| | 7.92 | 45.877 | 11.657 |
| 12 | -0.03 | 30.852 | 8.260 |
| | 2.25 | 70.914 | 17.969 |
| | 4.25 | 47.960 | 12.786 |
| | 6.13 | 40.304 | 10.379 |
| | 8.00 | 35.450 | 9.563 |
| 13 | -0.10 | 68.263 | 14.656 |
| | 1.07 | 98.623 | 21.050 |
| | 2.08 | 122.983 | 28.116 |
| | 4.02 | 88.581 | 19.227 |
| | 6.10 | 77.589 | 16.771 |
| | 8.10 | 69.466 | 15.085 |
| 14 | 1.02 | 66.823 | 13.196 |
| | 2.43 | 75.367 | 14.827 |
| | 4.02 | 63.294 | 12.060 |
| | 6.10 | 48.993 | 9.059 |
| | 8.02 | 35.207 | 5.852 |
| | -0.62 | 36.211 | 5.340 |
| | 1.12 | 97.037 | 17.224 |
| 15 | -1.75 | 31.124 | 5.997 |
| | 0.83 | 33.864 | 6.882 |
| | 1.92 | 61.286 | 13.123 |
| | 4.00 | 29.411 | 5.797 |
| | 5.90 | 22.595 | 4.390 |
| | 7.10 | 19.758 | 3.679 |
| 16 | 1.97 | 59.388 | 8.903 |
| | 5.33 | 51.557 | 7.009 |
| 17 | 2.03 | 95.156 | 16.796 |
| | 4.03 | 41.400 | 5.188 |
| | 5.95 | 23.634 | 2.358 |
| | 8.03 | 12.392 | 0.994 |
| 18 | 5.47 | 47.534 | 11.478 |

| | 7.87 | 32.785 | 8.997 |
|----|-------|---------|--------|
| 19 | -0.97 | 88.724 | 14.151 |
| | 1.20 | 158.668 | 30.242 |
| | 3.20 | 128.146 | 21.859 |
| | 5.20 | 100.281 | 15.687 |
| | 7.20 | 76.658 | 10.822 |
| 20 | -0.08 | 29.811 | 2.762 |
| | 2.42 | 80.068 | 11.926 |
| | 4.25 | 46.112 | 5.162 |
| | 6.08 | 33.278 | 3.229 |
| | 8.13 | 21.301 | 1.792 |